CLINICAL TRIAL: NCT05125198
Title: Translation, Cultural Adaptation, and Validation of Urdu Version of Victorian Institute of Sports Assessment - Achilles (VISA-A) Questionnaire for Athletes With Achilles Tendinopathy
Brief Title: Translation, Cultural Adaptation and Validation of Urdu Version of VISA-A Questionnaire
Acronym: VISA-A
Status: Completed | Type: Observational
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Sana Akram, Assistant Professor (University Institute of Physical Therapy), University of Lahore
Other Study IDs: ULahore
Record Dates: First submitted 2021-10-15; First posted 2021-11-18 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Achilles Tendinopathy
Keywords: Achilles tendinopathy; Validity; Reliability; Translation; VISA-A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to translate and validate the VISA-A questionnaire to the Urdu language, to interpret its psychometric properties, and to determine the reliability of scores obtained from the population of Pakistan. The translated version of the gold standard tool will be used by the local population as well as Urdu-speaking immigrants across the globe to better understand and report the severity of their symptoms. Hence, to improve quality of life across cultures, there is a need of standard outcome measures in Urdu language.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged over 18 years and both genders.
* Athletic population with the diagnosis of unilateral mid-portion or insertional Achilles tendinopathy, paratendinosis, partial tendon rupture with or without retrocalcaneal bursitis.
* With positive Painful arc sign and Royal London Hospital Test.
* Healthy individuals.

Exclusion Criteria:

* Complete rupture of Achilles tendon,
* Pregnant women and those with any history of radicular pain or lower extremity injury
* Previous surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Using the rule of Thumb: Minimum of 3 per items.
  * Total items in the questionnaire=8
  * As per rule of Thumb=8*5=40
  * n=40
  * *For better accuracy investigators will take sample size of 40 individuals with Achilles tendinopathy and 40 healthy ankles (Conventional group to assess known group validity).
  * So n=80
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change being assessed in interpretation of Severity of Achilles tendinopathy.among participants using translated version of VISA-A questionnaire. | 1 week
  VISA-A is consisted of eight questions that measured the domains of pain, function in daily living, and sporting activity. Results range from 0 to 100, where 100 represents the perfect score

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided